CLINICAL TRIAL: NCT03061123
Title: Patient Perceptions and Physician Assessment of Benefits and Risks of Oral Anticoagulation Due to Non-valvular Atrial Fibrillation
Brief Title: Patient Perceptions and Physician Assessment of Benefits and Risks of Oral Anticoagulation Due to Non-valvular AF
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 28-004 ex 15/16
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Health Literacy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
The risk of stroke is markedly elevated in patients with atrial fibrillation (AF). Oral anticoagulation (OAC) is indicated in individuals with moderate and high risk of stroke to the disadvantage of an increased burden from bleeding. Adequate knowledge of this disorder and understanding the benefits and hazards of antithrombotic treatment are essential to incorporate patient´s values and preferences in these decisions. This will further improve acceptance of recommended therapy and augment compliance with OAC.

The objective of this investigation is to compare patient´s perceptions and physician´s assessments of benefits and risks of OAC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and ECG-documented non-valvular atrial fibrillation
* New indication for oral anticoagulation (OAC)
* Ability of informed consent

Exclusion Criteria:

* Existing OAC therapy
* Valvular heart disease
* History of valve surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation with new indication for anticoagulation.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Comparison of subjective stroke risk perception with CHA2DS2-VASc score | Baseline
Comparison of subjective bleeding risk perception with HAS-BLED score | Baseline

SECONDARY OUTCOMES:
Relationship between accurate perception of stroke and bleeding risks and baseline parameters (highest completed level of education, subjective level of information) | Baseline

CONTACTS AND LOCATIONS:
Locations (8):
- Austria (8):
  - LKH Feldbach, Feldbach
  - LKH Fürstenfeld, Fürstenfeld
  - Hospital Barmherzige Brueder Eggenberg, Graz
  - Hospital Barmherzige Brueder Marschallgasse, Graz
  - Hospital Elisabethinen, Graz
  - Medical University of Graz, Graz
  - LKH Hartberg, Hartberg
  - Ordination Dr. Zweiker, Straden

REFERENCES:
- [Derived] Zweiker D, Zweiker R, Winkler E, Roesch K, Schumacher M, Stepan V, Krippl P, Bauer N, Heine M, Reicht G, Zweiker G, Sprenger M, Watzinger N. Association between subjective risk perception and objective risk estimation in patients with atrial fibrillation: a cross-sectional study. BMJ Open. 2017 Sep 25;7(9):e018242. doi: 10.1136/bmjopen-2017-018242. PMID 28951417